CLINICAL TRIAL: NCT00969501
Title: Investigator Initiated, Exploratory Case Study Three Injections of EUFLEXXA (Sodium Hyaluronate)Treatment of Chronic Shoulder Pain Associated With Osteoarthritis
Brief Title: Three Injections of EUFLEXXA (Sodium Hyaluronate) for Treatment of Chronic Shoulder Pain Associated With Osteoarthritis (OA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia Institute for Clinical Research, LLC (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Arnold J. Weil, M.D., M.D./CEO/Principal Investigator, Georgia Institute for Clinical Research, LLC
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EUF-SHO-0001
Record Dates: First submitted 2009-08-31; First posted 2009-09-01 (Estimated); Results first posted 2013-05-07 (Estimated); Last update posted 2013-05-07 (Estimated); Status verified 2013-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EUFLEXXA (Experimental): ACTIVE CONTROL
  Interventions: Drug: EUFLEXXA

INTERVENTIONS:
Drug: EUFLEXXA — 2.5 mL of EUFLEXXA (per injection) x 3 injections

SUMMARY:
The hypothesis of this study is that by using 3 injections of EUFLEXXA, there will be an improvement in pain levels and range of motion.

DETAILED DESCRIPTION:
To demonstrate that EUFLEXXA is safe for the treatment of chronic shoulder pain associated with osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Be age 30 to 79
2. Give written informed consent for trial participation
3. Must have shoulder pain for a minimum of 6 months but less than 5 years
4. Must have a Pain Intensity Score of > 5
5. Must be willing to discontinue all pain medications 24 hours prior to each clinic visit
6. Must have a stable pain medication regime 1 month prior to treatment
7. Agrees to maintain pain medication doses within 30% (increase or decrease) of the Baseline dose

Exclusion Criteria:

1. Any history of full thickness rotator cuff tear or joint effusion
2. A diagnosis of chronic acromioclavical disease, active epicondylitis, or active Carpal Tunnel Disease
3. Has had more than 2 corticosteroid injections in the previous 3 months
4. Has an infection or an inflammatory condition of the trial shoulder
5. Has acute or inflammatory arthropathy in the trial shoulder, e.g. gouty arthritis, psoriatic arthritis or rheumatoid arthritis. Has a history of systemic inflammatory arthropathies, e.g. polyarthritis, rheumatoid arthritis, psoriatic arthritis or gout
6. Has severe joint effusion of the trial shoulder
7. Has a diagnosis of cancer within the past 5 years (basal cell carcinoma is not excluded)
8. Has had any hyaluronate agent or other chondroprotective agents in the trial shoulder
9. Has a hypersensitivity to HA products, eggs, birds or feathers
10. Has a history of substance abuse, alcohol abuse or psychiatric condition, that in the opinion of the Investigator, will potentially interfere with participation
11. Has any medical condition that may increase the risk associated with intra-articular injections, to include (but are not limited to): thrombocytopenia, blood disorders treated with warfarin or anticoagulants, anemia or other concomitant diseases that, in the opinion of the Investigator, will interfere with the evaluation of the trial treatment, e.g., renal or liver disease, uncontrolled diabetes, significant cardiovascular, immune deficiency, or infectious disease
12. Is actively involved in a litigation involving Workers' Compensation
13. Is a female that is pregnant, planning to become pregnant or is lactating
14. Has participated in a clinical trial within the past four weeks

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arnold J. Weil, M.D., Principal Investigator — Georgia Institute for Clinical Research, LLC
Locations (1):
- Georgia Institute for Clinical Research, LLC, Marietta, Georgia, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- EUFLEXXA: All subjects received three injections (one each, in weeks 0 [baseline], 1, and 2 of high molecular weight hyaluronate (2.5 mL each) using standard injection techniques in the anterior or posterior approach. Sub- jects were evaluated at screening and baseline, and at weeks 1, 2, 6, 14, 26, and 27 (last evaluation by telephone).
Period: Overall Study
Arm/Group | EUFLEXXA
Started | 32
Completed | 27
Not Completed | 5

BASELINE CHARACTERISTICS:
Arm/Group | EUFLEXXA
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 31
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 59.1 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 16
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Reduction in Pain by the Scores.
Description: Greater than 50 percent reduction in pain scores from baseline.
Time Frame: 6 months
Population: ￼
Measure: Number; unit: participants
Arm/Group | EUFLEXXA
Number analyzed (Participants) | 27
participants | 25

ADVERSE EVENTS:
Arm/Group | EUFLEXXA
Serious Adverse Events (participants affected / at risk) | 0/32
Other Adverse Events (participants affected / at risk) | 0/32

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No